CLINICAL TRIAL: NCT03684187
Title: Mindfulness - Based Intervention in the Treatment of Fatigue in Patients With Primary Biliary Cholangitis: A Pilot Study
Brief Title: Mindfulness - Based Intervention in the Treatment of Fatigue in Patients With Primary Biliary Cholangitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit and change in funding status.
Sponsor: Yale University (Other)
Collaborators: American Liver Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000022299
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress in Control for Healthy Liver (SynC-HL) Intervention: (Experimental): This mindfulness based intervention to target healthy liver focuses on teaching skills of mindfulness, yoga and self-control to improve lifestyle choices and decision making.
  Interventions: Behavioral: Mindfulness Based Intervention

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — Mindfulness - Based Intervention (MBI) Course:
  The 8-week MBI program is comprised of an orientation session, 8 separate weekly sessions of 2.5 hours and also a 7.5 hour retreat session on a weekend day. The orientation session will include an introductory session, description of the course and will include completion of stress surveys. During the orientation session, there will be explanation to the patients of objectively the basis of mindfulness teaching. The role of the stress surveys that are conducted are to assess an individual's degree of stress prior to the initiation of any mindfulness practice teaching.
  Subjects will also be asked to wear a BodyGuard 2 (BG2) for parts of the study, on average of 7 days at baseline, end of the control phase, end of intervention phase, and end of 48 week follow up period. This will track subjects heart rate (HR), HR variability, VO2, energy expenditure and activity.

SUMMARY:
To assess the efficacy of mindfulness-based intervention (MBI) intervention in the treatment of moderate or severe fatigue in patients with primary biliary cholangitis (PBC).

DETAILED DESCRIPTION:
Aim 1: To assess the efficacy of mindfulness-based intervention (MBI) in the treatment of moderate or severe fatigue in patients with primary biliary cholangitis (PBC).

Hypothesis: MBI is feasible in PBC patients with fatigue and will result in improvement in symptoms of fatigue.

Aim 2: To assess the impact of MBI in physical activity levels, daytime somnolence, autonomic symptoms, functional status, cognitive dysfunction and anxiety and depressive symptoms of patients with PBC with moderate or severe fatigue.

Hypothesis: MBI will result in an improvement in physical activity levels, daytime somnolence, autonomic symptoms, functional status, cognitive dysfunction and anxiety and depressive symptoms in patients with PBC who have moderate or severe fatigue.

Aim 3: To evaluate the effects of MBI on candidate markers and/or cytokines of fatigue and physiological stress, including hepatic panel, antimitochondrial (AMA) titers, IL-1β, IL-6, TNFα, cortisol, leptin, CRP, BDNF, MIF, and CD74 levels and other relevant markers.

Hypothesis: MBI will result in a decrease of levels of above mentioned markers of fatigue and physiological stress in patients with PBC who have moderate or severe fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Primary Biliary Cholangitis as defined by previously published criteria
* On stable therapy with UDCA for at least 6 months before enrollment
* Primary Biliary Cholangitis-40 fatigue domain score > 33
* The ability to provide written consent

Exclusion Criteria:

* A known medical condition or metabolic disorder sufficient to explain fatigue such as anemia, thyroid disease, renal failure, use of beta-blockers and untreated depression
* Active drug or alcohol use or history of drug and/or stimulant abuse
* History of psychosis
* Modification of treatment for underlying PBC in the preceding six months
* Other serious coexistent conditions such as pre-existing advanced malignancy or severe cardiopulmonary disease which would be expected to limit their life expectancy
* Anticipated need for transplantation in one year (Mayo survival model <80% one-year survival without transplant) or MELD above 15
* Recurrent variceal bleeding, presence of diuretic-resistant ascites, or spontaneous encephalopathy
* Non-proficiency in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Change in fatigue severity | 16 weeks
  Change in fatigue severity, assessed by the fatigue domain of the Primary Biliary Cholangitis-40 (PBC-40) questionnaire, of greater than 5 units at 16 weeks (end of MBI program) compared to baseline

SECONDARY OUTCOMES:
Change in fatigue severity | 8 weeks
  Change in fatigue severity, assessed by the fatigue domain of the Primary Biliary Cholangitis-40 (PBC-40) questionnaire of greater than 5 units compared to baseline.
Change in fatigue severity | 24 weeks
  Change in fatigue severity, assessed by the fatigue domain of the Primary Biliary Cholangitis-40 (PBC-40) questionnaire of greater than 5 units compared to baseline.
Change in fatigue severity | 36 weeks
  Change in fatigue severity, assessed by the fatigue domain of the Primary Biliary Cholangitis-40 (PBC-40) questionnaire of greater than 5 units compared to baseline.
Change in fatigue severity | 48 weeks
  Change in fatigue severity, assessed by the fatigue domain of the Primary Biliary Cholangitis-40 (PBC-40) questionnaire of greater than 5 units compared to baseline.
Change in measurements of physical activity | 2 weeks
  Change in measurements of physical activity, measured by BodyGuard compared to baseline.
Change in measurements of physical activity | 8 weeks
  Change in measurements of physical activity, measured by BodyGuard compared to baseline.
Change in measurements of physical activity | 16 weeks
  Change in measurements of physical activity, measured by BodyGuard compared to baseline.
Change in measurements of physical activity | 48 weeks
  Change in measurements of physical activity, measured by BodyGuard compared to baseline.
Change in daytime somnolence | 8 weeks
  Change in daytime somnolence, assessed using the Epworth Sleepiness Scale (ESS) compared to baseline.
Change in daytime somnolence | 16 weeks
  Change in daytime somnolence, assessed using the Epworth Sleepiness Scale (ESS) compared to baseline.
Change in daytime somnolence | 24 weeks
  Change in daytime somnolence, assessed using the Epworth Sleepiness Scale (ESS) compared to baseline.
Change in daytime somnolence | 36 weeks
  Change in daytime somnolence, assessed using the Epworth Sleepiness Scale (ESS) compared to baseline.
Change in daytime somnolence | 48 weeks
  Change in daytime somnolence, assessed using the Epworth Sleepiness Scale (ESS) compared to baseline.
Change in vasomotor autonomic symptoms | 8 weeks
  Change in vasomotor autonomic symptoms assessed by the Orthostatic Grading Scale (OGS) compared to baseline.
Change in vasomotor autonomic symptoms | 16 weeks
  Change in vasomotor autonomic symptoms assessed by the Orthostatic Grading Scale (OGS) compared to baseline.
Change in vasomotor autonomic symptoms | 24 weeks
  Change in vasomotor autonomic symptoms assessed by the Orthostatic Grading Scale (OGS) compared to baseline.
Change in vasomotor autonomic symptoms | 36 weeks
  Change in vasomotor autonomic symptoms assessed by the Orthostatic Grading Scale (OGS) compared to baseline.
Change in vasomotor autonomic symptoms | 48 weeks
  Change in vasomotor autonomic symptoms assessed by the Orthostatic Grading Scale (OGS) compared to baseline.
Change in functional status | 8 weeks
  Change in functional status assessed by the Patient-Reported Outcomes Measurement Information System Health Assessment Questionnaire (PROMIS HAQ) compared to baseline.
Change in functional status | 16 weeks
  Change in functional status assessed by the Patient-Reported Outcomes Measurement Information System Health Assessment Questionnaire (PROMIS HAQ) compared to baseline.
Change in functional status | 24 weeks
  Change in functional status assessed by the Patient-Reported Outcomes Measurement Information System Health Assessment Questionnaire (PROMIS HAQ) compared to baseline.
Change in functional status | 36 weeks
  Change in functional status assessed by the Patient-Reported Outcomes Measurement Information System Health Assessment Questionnaire (PROMIS HAQ) compared to baseline.
Improvement in functional status | 48 weeks
  Improvement in functional status assessed by the Patient-Reported Outcomes Measurement Information System Health Assessment Questionnaire (PROMIS HAQ) compared to baseline.
Change in cognitive dysfunction | 8 weeks
  Change in cognitive dysfunction assessed by the Cognitives Failures (COGFAIL) questionnaire compared to baseline.
Change in cognitive dysfunction | 16 weeks
  Change in cognitive dysfunction assessed by the Cognitives Failures (COGFAIL) questionnaire compared to baseline.
Change in cognitive dysfunction | 24 weeks
  Change in cognitive dysfunction assessed by the Cognitives Failures (COGFAIL) questionnaire compared to baseline.
Change in cognitive dysfunction | 36 weeks
  Change in cognitive dysfunction assessed by the Cognitives Failures (COGFAIL) questionnaire compared to baseline.
Change in cognitive dysfunction | 48 weeks
  Change in cognitive dysfunction assessed by the Cognitives Failures (COGFAIL) questionnaire compared to baseline.
Change in anxiety and depressive symptoms | 8 weeks
  Change in anxiety and depressive symptoms assessed by the Hospital Anxiety and Depression Scale (HADS) compared to baseline.
Change in anxiety and depressive symptoms | 16 weeks
  Change in anxiety and depressive symptoms assessed by the Hospital Anxiety and Depression Scale (HADS) compared to baseline.
Change in anxiety and depressive symptoms | 24 weeks
  Change in anxiety and depressive symptoms assessed by the Hospital Anxiety and Depression Scale (HADS) compared to baseline.
Change in anxiety and depressive symptoms | 36 weeks
  Change in anxiety and depressive symptoms assessed by the Hospital Anxiety and Depression Scale (HADS) compared to baseline.
Change in anxiety and depressive symptoms | 48 weeks
  Change in anxiety and depressive symptoms assessed by the Hospital Anxiety and Depression Scale (HADS) compared to baseline.
Change in overall health status | 8 weeks
  Change in overall health status, assessed by the Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) compared to baseline.
Change in overall health status | 16 weeks
  Change in overall health status, assessed by the Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) compared to baseline.
Change in overall health status | 24 weeks
  Change in overall health status, assessed by the Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) compared to baseline.
Change in overall health status | 36 weeks
  Change in overall health status, assessed by the Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) compared to baseline.
Change in overall health status | 48 weeks
  Change in overall health status, assessed by the Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) compared to baseline.

OTHER OUTCOMES:
Changes in anti-mitochondria antibody (AMA) titers | 8 weeks
  Changes in anti-mitochondria antibody (AMA) titers, IL-1β, IL-6, TNFα, leptin, cortisol, CRP, BDNF, MIF, CD74 levels and other pertinent biomarkers, compared to baseline.
Changes in anti-mitochondria antibody (AMA) titers | 16 weeks
  Changes in anti-mitochondria antibody (AMA) titers, IL-1β, IL-6, TNFα, leptin, cortisol, CRP, BDNF, MIF, CD74 levels and other pertinent biomarkers, compared to baseline.
Changes in anti-mitochondria antibody (AMA) titers | 48 weeks
  Changes in anti-mitochondria antibody (AMA) titers, IL-1β, IL-6, TNFα, leptin, cortisol, CRP, BDNF, MIF, CD74 levels and other pertinent biomarkers, compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Silveira, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine - Digestive Diseases, New Haven, Connecticut, United States